CLINICAL TRIAL: NCT03825835
Title: Does the Use of Higher Versus Lower Oxygen Concentration Improve Neurodevelopmental Outcomes at 18-24 Months in Very Low Birthweight Infants - The HiLo-Trial
Brief Title: 30% or 60% Oxygen at Birth to Improve Neurodevelopmental Outcomes in Very Low Birthweight Infants
Acronym: HiLo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Toronto (Other); University of Sydney (Other); Dalhousie University (Other); McMaster University (Other); University of Manitoba (Other); McGill University (Other); University of Calgary (Other); Memorial University of Newfoundland (Other); University College Cork (Other); University of British Columbia (Other); Laval University (Other); Université de Montréal (Other); University of Ottawa (Other); Queen's University (Other); Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00083931
Record Dates: First submitted 2019-01-25; First posted 2019-01-31 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Premature Infant; Respiratory Distress Syndrome in Premature Infant; Neurodevelopmental Outcome
Keywords: Delivery Room; Resuscitation; Premature Infant; Oxygen
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessed will be unaware of group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30% group (Active Comparator): Infants in the 30% oxygen group will remain in 30% oxygen (O2) until 5 min of age. At 5 min of age, the clinical team will assess oxygen saturation (SpO2). If SpO2 is <85%, O2 should be increased by 10-20% every 60 sec to achieve SpO2 of 85% or greater or a SpO2 of 90-95% at 10 min of age. If SpO2 are greater than 95% at or before 5 min of age, O2 should be decreased stepwise (every 60 sec) with an aim to maintain SpO2 of 85% or greater during 5-10 min of age or 90-95% at and beyond 10 min of age.
  Intervention: Infants randomized to the 30% oxygen group will receive 30% oxygen at birth for the first 5 minutes. At 5 minutes oxygen can be adjusted as needed.
  Interventions: Drug: 30% oxygen group
- 60% group (Experimental): Infants in the 60% oxygen group will remain in 60% oxygen (O2) until 5 min of age. At 5 min of age, the clinical team will assess oxygen saturation (SpO2). If SpO2 is <85%, O2 should be increased by 10-20% every 60 sec to achieve SpO2 of 85% or greater or a SpO2 of 90-95% at 10 min of age. If SpO2 are greater than 95% at or before 5 min of age, O2 should be decreased stepwise (every 60 sec) with an aim to maintain SpO2 of 85% or greater during 5-10 min of age or 90-95% at and beyond 10 min of age.
  Intervention: Infants randomized to the 60% oxygen group will receive 60% oxygen at birth for the first 5 minutes. At 5 minutes oxygen can be adjusted as needed.
  Interventions: Drug: 60% oxygen group

INTERVENTIONS:
Drug: 30% oxygen group — Infants in the 30% oxygen group will remain in 30% oxygen (O2) until 5 min of age. At 5 min of age, the clinical team will assess oxygen saturation (SpO2). If SpO2 is <85%, O2 should be increased by 10-20% every 60 sec to achieve SpO2 of 85% or greater or a SpO2 of 90-95% at 10 min of age. If SpO2 are greater than 95% at or before 5 min of age, O2 should be decreased stepwise (every 60 sec) with an aim to maintain SpO2 of 85% or greater during 5-10 min of age or 90-95% at and beyond 10 min of age.
  Intervention: Infants randomized to the 30% oxygen group will receive 30% oxygen at birth for the first 5 minutes. At 5 minutes oxygen can be adjusted as needed.
  Arms: 30% group
Drug: 60% oxygen group — Infants in the 60% oxygen group will remain in 60% oxygen (O2) until 5 min of age. At 5 min of age, the clinical team will assess oxygen saturation (SpO2). If SpO2 is <85%, O2 should be increased by 10-20% every 60 sec to achieve SpO2 of 85% or greater or a SpO2 of 90-95% at 10 min of age. If SpO2 are greater than 95% at or before 5 min of age, O2 should be decreased stepwise (every 60 sec) with an aim to maintain SpO2 of 85% or greater during 5-10 min of age or 90-95% at and beyond 10 min of age.
  Intervention: Infants randomized to the 60% oxygen group will receive 60% oxygen at birth for the first 5 minutes. At 5 minutes oxygen can be adjusted as needed.
  Arms: 60% group

SUMMARY:
Preterm birth, or birth before 37 weeks' gestation, is increasingly common, occurring in 8 percent of pregnancies in Canada. Preterm birth is associated with many health complications, particularly when the birth happens before 29 weeks' gestation. At this gestational age, the lungs are not fully developed and it is not uncommon for infants to have problems breathing at the time of birth. One complication that can arise is when an infant stops breathing and needs to be resuscitated. When preterm babies need to be resuscitated doctors must take special care because of the small infant size and the immaturity of the brain and lungs. Oxygen is used to resuscitate babies who need it, but unfortunately there is disagreement about the best oxygen concentration to use. Oxygen concentration is important because both too much and too little oxygen can cause brain injury. This research aims to fill this knowledge gap by participating in an international clinical trial to compare the effects of resuscitating babies less than 29 weeks' gestational age with either a low oxygen concentration or a high oxygen concentration. The oxygen concentrations have been selected using the best available knowledge.

This will be a cluster randomized trial where each participating hospital will be randomized to either 30 or 60 percent oxygen for the recruitment of 30 infants, and afterwards randomized to the other group for the recruitment of another 30 infants. After the trial, the investigator will determine whether the babies resuscitated with low oxygen or those resuscitated with high oxygen have better survival and long-term health outcomes. This research fills a critical knowledge gap in the care of extremely preterm babies and will impact their survival both here in Canada and internationally.

DETAILED DESCRIPTION:
Purpose: Over the last 10 years, recommendations regarding the ideal level of oxygen for resuscitation in preterm infants have changed from 100 percent, down to low levels of oxygen (<30 percent), up to moderate concentration (30-65 percent). In addition, in 2010, oxygen saturation targeting was recommended as standard of care and this contributed to a change in clinical practice as clinicians were more likely and comfortable to start resuscitation at either 21percent (room air) or titrated levels of oxygen such as 30-40 percent. When the guidelines were again revised in 2015, the International Liaison Committee on Resuscitation (ILCOR) acknowledged that a critical knowledge gap continued to exist for the resuscitation of the preterm infants <37 weeks, highlighting the need to provide more concrete guidelines. This leaves clinicians in a challenging position. Despite the advances that have been achieved in perinatal and neonatal care, neonates are still vulnerable to the consequences of the oxidative effects from hyperoxia as well as the deleterious effects from hypoxia. A large, multi-centre international trial of sufficient sample size that is powered to look at safety outcomes such as mortality and adverse neurodevelopmental outcomes is required to provide the necessary evidenced to guide clinical practice with confidence.

Hypothesis: the null hypothesis for this study is that the incidence of mortality or abnormal neurodevelopmental outcomes at 24+/- 6 months corrected age will be no different by using either higher initial oxygen concentration of 60 percent compared to using lower initial oxygen concentration of 30 percent for resuscitation of preterm infants of 23 0/7- 28 6/7 weeks gestation.

Justification:

The use of supplementary oxygen may be crucial, but also potentially detrimental to premature infants at birth. High oxygen levels may lead to organ damage through oxidative stress, while low oxygen levels may lead to increased mortality. Excess oxygen exposure during the early post-birth period is associated with many complications and morbidities of preterm birth. Preterm infants have lower levels of anti-oxidant pathways consistent with their expected fetal environment of low oxygen exposure. Excess of oxygen free-radicals in infants intrinsically deficient in enzymatic antioxidants and non-enzymatic antioxidants may contribute to these morbidities. Pulmonary oxygen toxicity, through the generation of reactive oxygen and nitrogen species in excess of antioxidant defenses, is believed to be a major contributor to the development of bronchopulmonary dysplasia (BPD). Using lower oxygen concentrations at birth results in decreased oxidative stress markers and a decrease risk of developing BPD compared to higher oxygen concentrations. Other organs that may be damaged by such oxidative stress include kidneys, myocardium and the retina.

There is equally growing evidence that using lower oxygen concentrations will lead to lower oxygen saturation levels and bradycardia, which may lead to increased rates of mortality in this vulnerable group of infants. An individual patient analysis of clinical trials reported that 46% of preterm infants resuscitated with initial low oxygen concentration did not reach SpO2 of 80% at 5 min. This was associated with increased risk of major intraventricular hemorrhage (IVH), and an almost five times higher risk of death in this vulnerable group of infants. These data provide a warning note for the use of higher vs. lower initial oxygen concentration during delivery room resuscitation. As the investigator proceed in determining a safe range for resuscitation of ELBW/ELGA infants, it is highly likely that the optimum level of oxygen concentration is between the two extremes of 21 percent and 100 percent.

Objectives: To determine whether initial resuscitation of preterm neonates with 60 percent versus 30 percent oxygen results in better neurodevelopmental outcomes at 24+/- 6 months.

Research Method/Procedures: This will be a cluster crossover design, unmasked randomized controlled trial (RCT) comparing two oxygen concentrations at initiation of resuscitation. Infants will be placed on the resuscitation table with the initial steps of resuscitation carried out as per standard of care at each centre which usually follows current resuscitation guidelines. All centres will make every effort to establish adequate lung expansion using CPAP or positive pressure ventilation as needed. Enrolled infants will have a pulse oximeter sensor placed on the right arm in the first minute of life. Their resuscitation will be initiated with an oxygen concentration of 30 or 60 percent depending on the randomization sequence at the centre at the given time. Infants in the 30 percent group will remain in 30 percent oxygen until 5 min of age unless the infant's heart rate (HR) remains 100/min or less and does not show a tendency towards progressive increase before reaching 5 min of age or infant needs chest compression and/or epinephrine. No alteration in oxygen concentration will be made for an infant who is responding to resuscitation efforts with HR progressively increasing as minutes go by. At 5 min of age, the clinical team will assess oxygen saturation. If the saturation is less than 85 percent, oxygen should be increased by 10-20 percent every 60 sec to achieve saturations of 85 percent or greater or a saturation of 90-95 percent at 10 min of age. If saturations are greater than 95 percent at or before 5 min of age, oxygen should be decreased stepwise (every 60 sec) with an aim to maintain saturations of 85 percent or greater during 5-10 min of age or 90-95 percent at and beyond 10 min of age. The procedure for infants in the 60 percent group will be identical. The intervention duration for the trial will be the first 5 min after birth followed by initial monitoring/action for the next 5 min where titration in oxygen concentration will be made to achieve stability making a total of 10 min for study intervention. Titration of oxygen before 5 min after birth will only be made if the infant remains bradycardic (HR less than 100) and does not show a tendency towards a sustained increase in HR or if the oxygen saturation exceeds 95 percent. If the infant does not respond to ventilation with increasing HR in the first 5 min after birth, steps to ensure effective ventilation should be done before oxygen is titrated.

Plan for Data Analysis: Generalized linear mixed model with binary outcome and maximum likelihood estimate will be used to evaluate the effect of an oxygen concentration on the primary outcome (as a composite at 24+/- 6 months corrected age of all-cause mortality or the presence of a major neurodevelopmental outcome). To account for cluster crossover design of the study, effects of centers (clusters) and a period (oxygen concentration) within center will be considered random, and effects of a period (oxygen concentration) will be entered as a fixed effect. This hierarchical model allows for the correlation of patients within periods and within clusters. The model will be adjusted for gestational age and whether or not infant required mask ventilation as potential confounding variables. Similar generalized linear mixed models will be performed to evaluate the effect of group on secondary outcomes. In addition, three subgroup analysis will be performed: i) Gestational age will be categorized into 2 categories: 23+0- 25+6 vs. 26+0-28+6 weeks; ii) Breathing support will be categorized by infants supported only with CPAP vs. received mask ventilation; iii) Sex/Gender will be categorized into 2 categories: female vs. male. For subgroup analysis baseline characteristics will be compared using linear and generalized linear mixed models. Sensitivity analysis will be performed to analyze the missing data; however, a very low number of missing values are expected due to the design of the study.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at 23 0/7 weeks to 28 6/7 weeks' gestational age who will receive full resuscitation and are without major congenital abnormalities

Exclusion Criteria:

* Infants who are outborn - initial resuscitation not performed at the study centre
* Infants who are not born within the eligible gestational age range- this trial is specific to preterm infants
* Infants who are born with a major congenital abnormality- congenital abnormalities may affect oxygenation or neurodevelopmental outcomes
* Infants who will not receive full resuscitation at birth- these infants will not receive resuscitation

Ages: 0 Minutes to 10 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with composite outcome of all-cause mortality or the presence of a major neurodevelopmental outcomes | 24+/- 6 months corrected age
  Defined as any one of the following: Mortality or (i) cerebral palsy with an inability to walk unassisted; (ii) major developmental delay involving cognition or language; or (iii) visual (cannot fixate/legally blind, or corrected acuity < 6/60 in both eyes) or hearing impairment (requiring a hearing aid or cochlear implants).

SECONDARY OUTCOMES:
Number of intubation in the delivery room | first 15 minutes after birth
  Number of infants intubated in the delivery room
Death in the Neonatal Intensive Care Unit | During admission in the Neonatal Intensive Care Unit; no exact time frame can be given as this can happen after 1 day, 1 week, 1 months or up to 2-3 month. again deepening on gestational age and policy for transferring infants at participating centres.
  Number of infants died after admission in the Neonatal Intensive Care Unit
Number of participants who died in the delivery room | During resuscitation in the delivery room; for lay people: this time frame might be 10min or 1-3 hours, depending on the approaching each participating hospital
  Number of infants died in the delivery room during resuscitation
Number of participants with severe brain injury on cranial ultrasound | During NICU admission (up to 6 months)
  Severe grade 3 and 4 intraventricular or intraparenchymal hemorrhage according to Papile [44], periventricular leukomalacia, or ventriculomegaly based on neuroimaging studies (timing and frequency of imaging based on local site practices)
Number of participants with severe retinopathy of prematurity stage 3 or higher | During NICU admission (up to 6 months)
  As defined in the International Classification of ROP and/or ROP treated with laser, cryo-therapy, or intraocular injection therapy
Number of participants with necrotizing enterocolitis | During NICU admission (up to 6 months)
  Defined as modified Bell's criteria stage 2 or greater
Number of participants with hearing loss | 24+/- 6 months of age
  Audiometry will be performed to assess the presence or absence of severe hearing loss.
Number of participants with blindness | 24+/- 6 months of age
  Blindness will be defined as a corrected visual acuity of <20/200.
Number of participants with mortality | From birth up to 24+/- 6 months of age
  All cause mortality from birth until follow-up at 24+/- 6 months of age
Number of participants with cerebral palsy with an inability to walk unassisted | 24+/- 6 months of age
  Defined as cerebral palsy with an inability to walk unassisted
Number of participants with bronchopulmonary dysplasia at 36 weeks corrected age | At 36 weeks corrected age
  Defined as receiving any supplemental oxygen or any form of respiratory support (including invasive mechanical ventilation, non-invasive ventilation with continuous positive airway pressure, nasal intermittent positive pressure ventilation, or high-flow nasal cannula)
Number of participants with bronchopulmonary dysplasia at 40 weeks corrected age | At 40 weeks corrected age
  Defined as receiving any supplemental oxygen or any form of respiratory support (including invasive mechanical ventilation, non-invasive ventilation with continuous positive airway pressure, nasal intermittent positive pressure ventilation, or high-flow nasal cannula)
Total duration of mechanical ventilation via an endotracheal tube in days | Days during NICU Admission (up to 6 months)
  Days of receiving mechanical ventilation
Number of participants discharged home on oxygen | At NICU Discharge
  Infants who are discharged home with oxygen
Duration of any positive pressure respiratory support in days | Days during NICU Admission (up to 6 months)
  Defined as (invasive mechanical ventilation, non-invasive ventilation with continuous positive airway pres- sure, nasal intermittent positive pressure ventila- tion, or non-invasive neural assist ventilation or non-invasive high frequency ventilation, or high- flow nasal canula) in days
Duration of supplemental oxygen in days | Days during NICU Admission (up to 6 months)
  Number of days the infant receives any supplemental oxygen
Length of hospital stay in days | Days from birth to discharge (up to 6 months)
  number of days the infants I admitted in the nICU
Z-scores for weight, length, head circumference, and body mass index | At 36 weeks' corrected age
  we will calculate Z-scores for weight, length, head circumference, and body mass index
Differences in oxygen saturation in percentage | At 3, 5, and 10 min of age after birth
  we will compare the oxygen saturation in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmolzer, MD, PhD, Principal Investigator — University of Alberta
Locations (21):
- Canada (14):
  - Foothills Hospital, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - BC Children, Vancouver, British Colubia
  - Health Sciences, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - Newborn Health - IWK Health Centre, Halifax, Nova Scotia
  - Neonatal Intensive Care Unit - Hamilton Health Sciences, Hamilton, Ontario
  - Queen's University, Kingston, Ontario
  - CHEO, Ottawa, Ontario
  - Neonatal Intensive Care Unit - Mount Sinai Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill Univeristy, Montreal, Quebec
  - Chu University Laval, Québec, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec
- University College Cork, Cork, Ireland
- Spain (6):
  - Hospital Germans Tries i Pujol, Barcelona
  - Hospital Universitario Dexeus, Barcelona
  - Hospital de la Arrixaca, El Palmar
  - Hospital Las Palmas, Las Palmas de Gran Canaria
  - Hospital de Asturias, Oviedo
  - Hospital Universitario Materno Infantil Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
The data will be included in a prospectively planned IPD, which is called PROMOTION Other researchers can email the PI for more information at georg.schmoelzer@me.com
  Study protocol: https://link.springer.com/article/10.1186/s13063-024-08080-2
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after the publication of the primary results indefinitely
Access Criteria: Other researchers can email the PI for more information at georg.schmoelzer@me.com

REFERENCES:
- [Derived] Schmolzer GM, Asztalos EV, Beltempo M, Boix H, Dempsey E, El-Naggar W, Finer NN, Hudson JA, Mukerji A, Law BHY, Yaskina M, Shah PS, Sheta A, Soraisham A, Tarnow-Mordi W, Vento M; behalf of the HiLo trial collaborators. Does the use of higher versus lower oxygen concentration improve neurodevelopmental outcomes at 18-24 months in very low birthweight infants? Trials. 2024 Apr 4;25(1):237. doi: 10.1186/s13063-024-08080-2. PMID 38576007